CLINICAL TRIAL: NCT01625806
Title: A Single-Center, Open-Label, Parallel Study to Investigate the Effects of Multiple Doses of Ketoconazole on the Pharmacokinetics of a Single Oral Dose of RO4602522 in Healthy Male Subjects
Brief Title: A Study of The Effects of Multiple Doses of Ketoconazole on Single Dose Pharmacokinetics of RO4602522 in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: BP28236; 2012-001195-11 (EudraCT Number)
Record Dates: First submitted 2012-06-19; First posted 2012-06-21 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Healthy Volunteer
MeSH Terms: interventions — sembragiline; Ketoconazole

ARMS (2):
- RO4602522 (Active Comparator)
  Interventions: Drug: RO4602522
- RO4602522 + ketoconazole (Experimental)
  Interventions: Drug: RO4602522; Drug: ketoconazole

INTERVENTIONS:
Drug: RO4602522 — Single oral dose
Drug: ketoconazole — Multiple oral doses
  Arms: RO4602522 + ketoconazole

SUMMARY:
This single-center, open-label, parallel group study will evaluate the effects of multiple doses of ketoconazole on the pharmacokinetics of single oral dose RO4602522 in healthy male volunteers. All subjects will receive a single oral dose of RO4602522 on Day 1. Subjects assigned to Group 2 will additionally receive ketoconazole (200 mg orally every 12 hours) from Day 1 to Day 17.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects, 18 to 45 years of age, inclusive Healthy status is defined by absence of evidence of any active or chronic disease following detailed medical and surgical history and a complete physical examination
* Body mass index (BMI) 18 to 30 kg/m2 inclusive
* Male subjects and their partners of child-bearing potential must use two methods of contraception, one of which must be a barrier method, for the duration of the study and for 90 days after the last dose
* Non-smoker (not having smoked since at least 3 months prior to screening)

Exclusion Criteria:

* History of alcohol abuse or drug addiction (including soft drugs like cannabis products)
* Positive for hepatitis B, hepatitis C, or HIV infection
* Participation in an investigational drug or device study within 90 days prior to screening
* Concomitant disease or condition that could interfere with, or treatment of which might interfere with the conduct of the study, or that would, in the opinion of the investigator, pose an unacceptable risk to the subject in this study
* History of any disease or condition that could alter the absorption, metabolism or elimination of drugs
* Positive drug test and/or positive alcohol test
* Positive cotinine test
* Subject likely to need concomitant medication during the study period (including for dental conditions)
* Any confirmed significant allergic reactions against any drug, or multiple allergies in the judgment of the investigator

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2012-07; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Effect of multiple doses of ketoconazole on RO4602522 single dose pharmacokinetics: Area under the concentration-time curve (AUC) | Pre-dose and up to 10 hrs post-dose Day 1, and on Days 2-22

SECONDARY OUTCOMES:
Safety: Incidence of adverse events | approximately 3 months
RO4602522 metabolites: Plasma/urine concentrations | Pre-dose and up to 10 hrs post-dose Day 1, and on Days 2-22

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Zuidlaren, Netherlands